CLINICAL TRIAL: NCT00452582
Title: Phase 1 Study of Sildenafil (Viagra) Treatment of Subacute Ischemic Stroke
Brief Title: Sildenafil (Viagra) Treatment of Subacute Ischemic Stroke
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Failure to recruit in expected time period.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Brian Silver, MD, Henry Ford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HF-N-1
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; recovery; sildenafil
MeSH Terms: conditions — Ischemic Stroke | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): Orally administered sildenafil in addition to usual care.
  Interventions: Drug: Sildenafil (Viagra)
- Usual post-stroke care (Active Comparator): Usual post-stroke treatment including physical, occupational, and speech therapy.
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Sildenafil (Viagra) — Dose escalation (one of the following): 25 mg daily for 2 weeks, 50 mg daily for 2 weeks, 75 mg daily for 2 weeks, 50 mg twice daily for two weeks, 50 mg AM and 75 mg PM for 2 weeks, 75 mg twice daily for 2 weeks, 75 mg in AM and 100 mg in PM for 2 weeks, 100 mg twice daily for 2 weeks.
  Arms: Sildenafil
Other: Usual care — Physical therapy, occupational therapy, speech therapy
  Arms: Usual post-stroke care

SUMMARY:
Stroke is the third leading cause of death in the United States and the leading cause of serious long-term disability. Approximately 50% of the 750,000 people affected by stroke each year have residual physical impairment. Treatment options for recovery are limited at this time. Sildenafil (Viagra) has demonstrated the capability of significantly improving recovery in several animal experiments of stroke. This study is aiming to establish the safety of treatment with sildenafil in people with stroke with the ultimate aim of testing its usefulness to improve recovery.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the leading cause of serious long-term disability in the United States. Approximately 15-30% of stroke survivors are permanently disabled. Twenty eight percent of stroke patients are under age 65 which results in a loss of work income. While many restorative therapies are touted as promising for the treatment of ischemic stroke, to date none are approved for this purpose. Sildenafil (Viagra®), a phosphodiesterase type 5 inhibitor, has been shown to reduce mortality and improve the functional outcomes of young and aged rats when administered 24 hours and 7 days after stroke onset. Such results are encouraging and warrant further investigation in human stroke.

The specific aims of this study are to assess the safety of treating ischemic stroke patients with sildenafil (Viagra®) and to evaluate their outcomes at day 90. This will be a phase I dose-escalation study with cohort sizes of 12 patients (depending on the occurrence of serious adverse events). A total enrollment of 120 patients is planned. Patients who are between 4 and 7 days from stroke onset will receive 25, 50, 75, 100, 125, 150, 175, and 200 mg daily of sildenafil for a period of 14 days. Of the 120 patients, 24 will be randomly selected to receive standard treatment but will not receive sildenafil. All patients and physicians will be aware of treatment assignment. Evaluation of potential toxicity will be monitored throughout the course of treatment and during a formal visit at day 16 after initiation of treatment. Plasma monitoring of vascular endothelial growth factor (VEGF) will be made prior to treatment, at days 7, 16, 30, 60, and 90. Measurements of NIHSS scores, Rankin scores, and Barthel indices will be made at days 30, 60, and 90. Patients will also be assessed for color vision changes and sexual function during day 16 and day 90 visits. There will be every other day phone calls to patients while on treatment. The primary outcome measure will be death, recurrent stroke, and myocardial infarction during treatment. Exploratory analysis will include functional outcomes as measured on the neurological scales, and changes in VEGF levels in relation to clinical outcome.

The long-term objective is to identify a safe and easily administered treatment that improves functional outcome in patients with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke between 4 and 7 days after symptom onset.
* Patients age 18-80 years old.
* NIHSS score of 5-21 prior to treatment (within each cohort, there will be no more than 4 patients with NIHSS < 9 and no fewer than 4 patients with NIHSS > 11).
* Signed IRB-approved informed consent by patient or authorized representative.

Exclusion Criteria:

General:

* Participation in another study with an investigational drug or device.
* Women known to be pregnant, lactating, or of childbearing potential with a positive urine beta-HCG.
* Patients who cannot receive oral medications.
* Patients using sildenafil or other phosphodiesterase inhibitors within the previous 7 days of stroke.

Safety Related:

* Unstable angina.
* Myocardial infarction within 3 months.
* Current use of nitrate agents.
* Current use of alpha-channel antagonists.
* Current use of medications that inhibit the cytochrome p450 3A4 system. These medications include: amiodarone, aprepitant, bosentan, cimetidine, cisapride, clarithromycin, delavirdine, diltiazem, efavirenz, erythromycin, fluconazole, fluvoxamine, grapefruit juice, imatinib, itraconazole, ketoconazole,loratadine, mibefradil, mifepristone (RU-486), niacin, nefazodone, quinidine, quinine, ritonavir, saquinavir, tacrolimus, verapamil, voriconazole.
* St. John's Wort and phenytoin (inducers of cytochrome P450 3A4)
* Baseline systolic blood pressure less than 100 mmHg.
* Penile deformities.
* Creatinine > 1.5.
* Abnormal liver function studies.
* Patients with a previous history of sudden monocular vision loss Potentially Interfering with Outcomes Assessment:
* Prior history of dementia.
* Patients without fixed address or those deemed unlikely to present for follow-up by the investigator.
* Patients whose life expectancy is less than 90 days.
* Pre-stroke modified Rankin score > 2.
* Glucose greater than or equal to 400 mg/dL at presentation.
* Other serious illness (e.g., severe hepatic, cardiac, or renal failure; acute myocardial infarction; or a complex disease that may confound treatment assessment).
* Previous stroke or TIA within 30 days.
* Allergy or hypersensitivity to sildenafil or other phosphodiesterase inhibitors.
* History of sudden monocular visual disturbance.
* History of sudden unilateral hearing problem.

Imaging Related:

* Evidence of primary intraparenchymal hemorrhage on initial neuroimaging study.
* Neuroimaging evidence of nonvascular cause for the neurological symptoms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-04

PRIMARY OUTCOMES:
The maximum tolerated dose and toxicity profile of sildenafil treatment in patients with subacute ischemic stroke. | 2 weeks

SECONDARY OUTCOMES:
The estimated efficacy of sildenafil in comparison with concurrent patients randomized assigned to usual care. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian Silver, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Result] Silver B, McCarthy S, Lu M, Mitsias P, Russman AN, Katramados A, Morris DC, Lewandowski CA, Chopp M. Sildenafil treatment of subacute ischemic stroke: a safety study at 25-mg daily for 2 weeks. J Stroke Cerebrovasc Dis. 2009 Sep-Oct;18(5):381-3. doi: 10.1016/j.jstrokecerebrovasdis.2009.01.007. PMID 19717023